CLINICAL TRIAL: NCT02745366
Title: The Effect of Buccal Fat Pad Derived Mesenchymal Stem Cells Loaded on Allograft and Platelet-rich Plasma in Posterior Mandible Augmentation
Brief Title: Buccal Fat Pad Derived Stem Cells With Cortical Tenting in Posterior Mandible Reconstruction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arash Khojasteh, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbmu9217
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Alveolar Bone Loss; Atrophy
MeSH Terms: conditions — Alveolar Bone Loss; Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BFPSC+ (Experimental): The combination of BFPSC+FDBA+PRF is utilized in cortical tenting technique with block graft obtained from lateral ramus for posterior mandible augmentation procedure.
  Interventions: Procedure: BFPSC+FDBA+PRF
- BFPSC- (Active Comparator): The combination of FDBA+PRF is utilized in cortical tenting technique with block graft obtained from lateral ramus for posterior mandible augmentation procedure
  Interventions: Procedure: FDBA+PRF

INTERVENTIONS:
Procedure: BFPSC+FDBA+PRF
  Arms: BFPSC+
Procedure: FDBA+PRF
  Arms: BFPSC-

SUMMARY:
In this study the buccal fat pad derived stem cells (BFPSCs) is harvested from buccal fat pad tissue of the patients receiving posterior mandible augmentation. In the test group the patients receive a combination of platelet rich fibrin (PRF) and freeze dried bone allograft (FDBA) (SureOss, Hansbiomed, Korea) loaded with BFPSCs. The control group receivesFDBA (without any cells)+PRF. In all the groups the combination are placed between the recipient site and the block graft obtained from lateral ramus. The results will be evaluated by cone beam computed tomography (CBCT)and hematoxylin and eosin staining in 6 months.

DETAILED DESCRIPTION:
Autogenous bone blocks are harvested from lateral ramus.The buccal fat pad derived stem cells (BFPSCs) is harvested from buccal fat pad tissues. The BFPSCs will be loaded on freeze dried bone allograft (FDBA) (SureOss, Hansbiomed, Korea). Furthermore, twenty milliliters of the venous blood is obtained, placed and collected in a sterile tube, and centrifuged (GAC medical) for 14 minutes at 2800 rpm (approximately 400 g). Following centrifugation, three layers are separated in the tube: cellular plasma at the top, platelet rich fibrin (PRF) clot in the middle and red blood cells at the bottom of the tube. The PRF clot is separated by a sterile pincette.

The patients in the test group receives BFPSCs loaded on FDBA with PRF for posterior mandible augmentation and the control group receives combination of PRF and FDBA (lacking any cells). The BFPSCs+FDBA+PRF in the test group and FDBA+PRF in the control group are placed in the gap between the block graft and recipient site. The results will be evaluated by cone beam computed tomography (CBCT) in 6 months and microscopic evaluation of the biopsies by hematoxylin and eosine staining during implant placement.

ELIGIBILITY:
Inclusion Criteria:

* patients with posterior mandible edentulism and atrophic bone with less than 4mm bone width at bone crest or less than 8 mm bone height (considering 2-3 mm distance to anatomic structures)

Exclusion Criteria:

* smoking, history of malignancy, radiation, chemotherapy, pregnancy, systemic diseases contradicting dental and surgical treatments, conditions or drugs affecting bone remodeling or bone metabolism and connective tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
amount of regenerated bone | 6 months
  the amount of regenerated bone will be assessed by Image Pro software in CBCT images
amount of regenerated bone | 6 months
  the percent of regenerated bone will be assessed on bone biopsies obtained during implant insertion by H&E staining by microscope

CONTACTS AND LOCATIONS:
Overall Officials: Arash Khojasteh, DMD, OMFS, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- School of Dentristry at Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided